CLINICAL TRIAL: NCT02463708
Title: Evaluation of the PACE/PACENET BHL Caregiver Outreach and Telehealth Education Program
Brief Title: Evaluation of the PACE/PACENET BHL Caregiver Program
Acronym: CREST
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Magellan Health Services (Other)
Responsible Party: Principal Investigator, Mary Beth Gibbons, Ph.D., Director of Center for Psychotherapy Research. Professor of Psychiatry, Department of Psychiatry, Perelman School of Medicine, University of Pennsylvania
Other Study IDs: 819012
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Dementia
Keywords: Care Giver; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- BHL COTP Caregivers: Caregivers participate in the BHL COTP, which provides support, education, and care management services from a Behavioral Health Provider (BHP) in addition to the Telehealth Education Program (TEP), a manualized program that consists of various modules that seek to provide both education and psychosocial support for individuals caring for older adults with clinically significant cognitive impairment/dementia.
  Interventions: Behavioral: BHL COTP

INTERVENTIONS:
Behavioral: BHL COTP — The BHL COTP starts with an initial baseline assessment; following the baseline assessment, it is then divided into several core services. CG receive care management services, which includes contact, support, and active listening, as well as written material regarding caregiving and dementia and referral to appropriate community services. CGs also are offered the Telehealth Education Program (TEP) a manualized program developed to provide both education and psychosocial support for individuals caring for older adults with clinically significant cognitive impairment/dementia.

SUMMARY:
This project will conduct a retrospective clinical database review and a one-time research interview to evaluate outcomes among a sub-set of caregivers (CGs) who were enrolled in the Behavioral Health Laboratory (BHL) Caregiver Outreach and Telehealth Education Program (COTP). The investigators will recruit CGs whose Care Recipients (CR) met criteria for clinically significant cognitive impairment and/or dementia and who received care management services through the COTP.

DETAILED DESCRIPTION:
The University of Pennsylvania's Caregiver Resources, Education, & SupporT (CREST) Program seeks to improve the overall quality of life and wellbeing of older PACE/PACENET beneficiaries (or care recipients (CRs)) with cognitive impairment and their caregivers (CGs). Specifically, the program provides education, support, and services to both beneficiaries and CGs of PACE/PACENET beneficiaries who have filled a prescription for medication used to treat cognitive impairment. Many of these beneficiaries also meet criteria for clinically significant cognitive impairment/dementia. Thus, the level of contact and services varies as a function of reported needs and symptoms.

The CREST Program developed the BHL Caregiver Outreach and Telehealth Program (COTP) in an effort to address and minimize barriers to successful care management of a growing number of community-dwelling older adults. The COTP starts with an initial baseline assessment; following the baseline assessment, it is then divided into several core services. CGs receive care management services, which includes contact, support, and active listening, as well as written material regarding caregiving and dementia and referral to appropriate community services. CGs also are offered the Telehealth Education Program (TEP), a manualized program developed to provide both education and psychosocial support for individuals caring for older adults with clinically significant cognitive impairment/dementia.

This research project seeks to evaluate the feasibility, acceptability, and individual-level outcomes of a subset of participants engaged in the COPT program. Specifically, the investigators will examine the impact of the COPT program on the functioning and wellbeing of participating cognitively impaired PACE/PACENET beneficiaries and their informal CGs.

Retrospective clinical program data on COTP beneficiaries and the CGs collected at intake (i.e., baseline), over the course of care management, and at program termination (i.e., approximately 3 months following intake) will be extracted from clinical databases for program evaluation purposes. The researchers will use data collected during the clinical program to evaluate CR and CG characteristics, self-reported needs, care participation, and predictors of improved outcomes at 3 and 6 months.

A single follow-up research evaluation will be conducted at 6 months post baseline. This the 6 month follow-up research interviews will evaluate the extent to which a clinical care management program (COTP) for older adults with clinically significant cognitive impairment and/or dementia and the CGs, 1) facilitates access to and the use of medical and social services, and 2) improves CR (e.g., behavioral symptoms, delayed nursing home placement) and CG (e.g., CG mastery, burden, affect) outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and older, males and females.
2. The beneficiary screened positive for clinically significant cognitive impairment (BOMC score > 14) during the Care Recipient Baseline BHL COTP interview and agreed to allow COPT staff to speak with a CG, OR, the beneficiary could not complete the Care Recipient Baseline BHL COTP interview at all, agreed to allow COPT staff to speak with a CG on their behalf, and the CG verified that the beneficiary has clinically significant cognitive impairment (via AD8 score of 2 or more) and/or a dementia diagnosis made by a health care provider.
3. CG provides verbal informed consent to the use of retrospective clinical BHL COTP data and participation in the 6 Month Outcome Research Evaluation at the completion of the 3 Month Program Termination visit.

Exclusion Criteria:

* Not meeting the inclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caregivers of PACE/PACENET beneficiaries who are participating in the BHL COTP.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2013-11; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Revised Memory and Behavior Problems Checklist | 6 Months
  A checklist for dementia-related symptoms in 3 domains (memory impairment, depression, and disruptive behaviors) and associated CG burden.

SECONDARY OUTCOMES:
Lawton Caregiver Appraisal Scales | 6 Months
  A scale for caregiver satisfaction, mastery, demands, and perceived impact.
Desire to Institutionalize Scale | 6 Months
  A 6-item scale predictive of CGs actual institutionalization of care recipients.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Gibbons, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Department of Psychiatry (Center for Psychotherapy Research), University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wray LO, Shulan MD, Toseland RW, Freeman KE, Vasquez BE, Gao J. The effect of telephone support groups on costs of care for veterans with dementia. Gerontologist. 2010 Oct;50(5):623-31. doi: 10.1093/geront/gnq040. Epub 2010 May 27. PMID 20507926
- [Background] Mavandadi S, Patel S, Benson A, DiFilippo S, Streim J, Oslin D. Correlates of Caregiver Participation in a Brief, Community-Based Dementia Care Management Program. Gerontologist. 2017 Nov 10;57(6):1103-1112. doi: 10.1093/geront/gnw127. PMID 27927725
- [Background] Mavandadi S, Wray LO, DiFilippo S, Streim J, Oslin D. Evaluation of a Telephone-Delivered, Community-Based Collaborative Care Management Program for Caregivers of Older Adults with Dementia. Am J Geriatr Psychiatry. 2017 Sep;25(9):1019-1028. doi: 10.1016/j.jagp.2017.03.015. Epub 2017 Mar 27. PMID 28433550
- [Background] Mavandadi S, Wright EM, Graydon MM, Oslin DW, Wray LO. A randomized pilot trial of a telephone-based collaborative care management program for caregivers of individuals with dementia. Psychol Serv. 2017 Feb;14(1):102-111. doi: 10.1037/ser0000118. PMID 28134558
- [Derived] Gonzalez-Fraile E, Ballesteros J, Rueda JR, Santos-Zorrozua B, Sola I, McCleery J. Remotely delivered information, training and support for informal caregivers of people with dementia. Cochrane Database Syst Rev. 2021 Jan 4;1(1):CD006440. doi: 10.1002/14651858.CD006440.pub3. PMID 33417236